CLINICAL TRIAL: NCT07352930
Title: A Novel Intraoperative Fluorescence-guided System for Evaluating Margins During Breast-conserving Surgery for Breast Cancer: A Prospective Non-randomized Controlled Trial
Brief Title: A Novel Intraoperative Fluorescence-guided System for Evaluating Margins During Breast-conserving Surgery for Breast Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Kun Wang, Clinical Professor, Guangdong Provincial People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: KY2025-1339-01
Record Dates: First submitted 2026-01-13; First posted 2026-01-20 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Breast-Conserving Surgery
Keywords: Intraoperative Imaging; Fluorescence-Guided Surgery; Positive Margins
MeSH Terms: conditions — Margins of Excision | interventions — Drug Delivery Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EndoSCell Scanner (ES Scanner)-Assisted Intervention Group (Experimental): All enrolled participants will undergo the investigational intervention, which integrates the use of the EndoSCell Scanner (ES Scanner) system into the standard breast-conserving surgery (lumpectomy) procedure.
  Interventions: Device: EndoSCell Scanner (ES Scanner) System

INTERVENTIONS:
Device: EndoSCell Scanner (ES Scanner) System — The EndoSCell Scanner (ES Scanner) is an intraoperative fluorescence imaging system designed to provide real-time, cellular-level visualization of the surgical cavity walls during breast-conserving surgery (lumpectomy). The system consists of a handheld imaging probe connected to a console and display. During surgery, after removal of the main tumor specimen, the cavity walls are topically stained with fluorescein sodium and methylene blue. The ES Scanner probe is then placed against the tissue, where it uses blue light excitation to detect fluorescence patterns associated with residual cancer cells. The system processes and displays these images in real-time, highlighting areas suspected of containing residual carcinoma. This visual guidance is intended to assist the surgeon in precisely excising additional tissue margins ("therapeutic shaves") from specific, suspicious locations, to achieve a negative (cancer-free) surgical margin during the initial operation.

SUMMARY:
The goal of this clinical trial is to learn if a novel intraoperative fluorescence-guided system (EndoSCell Scanner) can help surgeons more accurately remove all cancerous tissue during breast-conserving surgery in female patients aged 18 years or older, with primary breast cancer. The main questions it aims to answer are:

* Does the use of the EndoSCell Scanner system lower the rate of secondary surgeries needed due to positive cancer margins after the initial operation?
* How accurate is the EndoSCell Scanner system in detecting residual cancer cells on the walls of the surgical cavity during the operation?

Researchers will compare the surgical outcomes using the EndoSCell Scanner guidance to the expected outcomes from standard surgical practice without this technology to see if the system is effective.

Participants will:

* Receive their planned breast-conserving surgery (lumpectomy).
* Have their surgical cavity scanned with the EndoSCell Scanner device after the main tumor is removed.
* Have additional tissue removed from the cavity wall if the scanner indicates a potential cancer residue.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically confirmed diagnosis of primary invasive breast cancer, ductal carcinoma in situ (DCIS), or invasive breast cancer with a DCIS component. Acceptable diagnostic methods include core needle biopsy or fine-needle aspiration biopsy.
2. Female, age ≥ 18 years.
3. Scheduled to undergo breast-conserving surgery (lumpectomy) for the malignant breast lesion.
4. Willing and able to comply with the study procedures and follow-up.
5. Has provided written informed consent.
6. No other uncontrolled serious medical conditions aside from the cancer diagnosis (see Exclusion Criteria for details).
7. Adequate organ and bone marrow function, defined as:

   * White blood cell count > 3,000/μL
   * Platelet count > 75,000/μL
   * Total bilirubin ≤ institutional upper limit of normal (ULN)
   * AST (SGOT) / ALT (SGPT) < 2.5 × institutional ULN
   * Serum creatinine ≤ 1.5 mg/dL, OR creatinine clearance > 60 mL/min/1.73 m² (for participants with serum creatinine levels above institutional ULN)
8. ECOG performance status of 0 or 1.

Exclusion Criteria:

1. Planned bilateral mastectomy.
2. Pregnancy or lactation.
3. Suspected pregnancy.
4. Use of any investigational drug within 30 days prior to enrollment.
5. Prior injection of ICG or other fluorescent dyes for sentinel lymph node mapping on the day of surgery, before the planned lumpectomy cavity scan with the study device.
6. Unresolved adverse events from previous medications or diagnostic agents.
7. Uncontrolled hypertension, defined as persistent systolic blood pressure > 180 mmHg or diastolic blood pressure > 110 mmHg. Patients with known hypertension must be stable on medication within these limits.
8. History of allergy to any oral or intravenous contrast agent.
9. Uncontrolled comorbidities, including but not limited to:

   * Active infection
   * Symptomatic congestive heart failure
   * Unstable angina pectoris
   * Cardiac arrhythmia
   * Hospitalization for COPD or asthma within the past 12 months
   * Psychiatric illness/social situations that would limit compliance with study requirements.
10. Any condition where, in the investigator's judgment, participation would not be in the best interest of the participant.
11. Planned re-excision lumpectomy due to positive margins from a prior surgery performed before enrollment.
12. Prior surgical history in the ipsilateral breast, including breast cancer surgery, mastectomy, breast reconstruction, or implant placement.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Reoperation Rate Due to Positive Surgical Margins | From the date of the initial lumpectomy (Day 0) until the receipt of the final postoperative pathology report and surgical decision, assessed up to 30 days post-surgery.
  The proportion of participants who undergo a secondary surgical procedure (re-excision or mastectomy) following the initial breast-conserving surgery, where the decision for reoperation is solely based on a final postoperative pathology report indicating a positive margin (invasive carcinoma at the inked surface or DCIS within 2 mm of the inked surface).
Diagnostic Accuracy (Sensitivity and Specificity) of the ES Scanner | Intraoperative. Assessment occurs during the surgical procedure, immediately following the ES Scanner imaging and the excision of any guided "therapeutic shave" margins. The outcome is calculated after all excised tissue has undergone final pathological
  The performance of the EndoSCell Scanner in correctly identifying the presence or absence of residual carcinoma on cavity walls during surgery, as determined by subsequent histopathological analysis. Sensitivity measures the proportion of truly positive margins correctly identified by the scanner. Specificity measures the proportion of truly negative margins correctly identified by the scanner.

SECONDARY OUTCOMES:
Mean Absolute Volume of Therapeutic Shave Tissue | Intraoperative. Measured immediately after tissue excision
  The average volume (in cubic centimeters, cc) of tissue excised as ES Scanner-guided Therapeutic Shaves (T-shaves) per participant. Volume calculation for each T-shave: length (cm) × width (cm) × depth (cm). The total T-shave volume per participant is the sum of all individual T-shave volumes. For participants who did not undergo T-shave excision, the volume is recorded as 0 cc.
Mean Proportion of Therapeutic Shave Volume to Total Resection Volume | Intraoperative. Calculated after all tissue from the initial surgery is measured
  The average percentage contribution of the T-shave volume to the total volume of all tissue resected during the initial surgery. Calculation: (T-shave volume) / (Main specimen volume + SOC shave volume + T-shave volume) × 100%.
Average Number of SOC Shaves and Therapeutic Shaves per Participant | Intraoperative. Recorded upon completion of the initial surgical procedure.
  The mean count of Standard of Care (SOC) shave margins and ES Scanner-guided Therapeutic Shave (T-shave) margins excised for each participant during the initial surgery.
Number of Participants Recommended for Secondary Surgery Due to Positive Margins | From surgery date until receipt of final pathology report and surgical recommendation, assessed up to 30 days post-initial surgery.
  The count of participants for whom a secondary surgery (re-excision or mastectomy) is recommended based on a final postoperative pathology report confirming positive margins on any initially resected specimen.
Detection Rate of Residual Carcinoma in Therapeutic Shaves | From the surgery date until receipt of the final pathology report for all initially excised tissue, assessed up to 30 days post-surgery.
  The proportion of participants in whom residual carcinoma (invasive or DCIS) is pathologically confirmed in at least one of the ES Scanner-guided therapeutic shave (T-shave) specimens excised during the initial surgery. Calculation: (Number of participants with positive T-shaves) / (Total number of participants) × 100%.
Proportion of Secondary Surgeries with Confirmed Residual Carcinoma | From the date of secondary surgery until receipt of its final pathology report, assessed up to 60 days post-initial surgery.
  Among participants who undergo a secondary surgery, the proportion in whom residual carcinoma is pathologically confirmed in the tissue specimens from that secondary procedure.
Record of Intraoperative Device Issues or Malfunctions | Intraoperative. Recorded in real-time during device use.
  The frequency, type, and impact (e.g., on data acquisition, procedural continuity) of any device problems, technical failures, or operational difficulties encountered with the ES Scanner system during surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong Provincial People's Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No